CLINICAL TRIAL: NCT05482997
Title: Athlete Whey Protein Sensitivity: Prevalence and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, Brittanie L. Lockard, Assistant Professor, University of the Incarnate Word
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-1154-EXP
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Food Intolerance
MeSH Terms: conditions — Food Intolerance | interventions — Whey

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blinded (subject only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group: Subjects with no protien intake (No Intervention): 20 subjects will receive no intervention for 10 weeks but complete performance tests and assessments during weeks 0, 4, 6, and 10.
- Whey Protein, Then Plant-based Protein (Experimental): Performance tests/assessments will be conducted as baseline testing without whey protein, followed by four weeks of whey protein intervention consisting of one 70cc (32g) scoop of supplement provided within an hour after athletic practice, five days a week. For athletes with more than one practice a day, the supplement will be provided after the strength training session. The powder will be shaken with 8-12oz water. Performance measured at the end of 4 weeks.
  After a two-week washout period, they will undergo another performance evaluation and begin the same protein supplement regimen, but with a 70cc (32g) scoop of the plant-based protein supplement.
  Interventions: Dietary Supplement: Whey Protein Concentrate; Dietary Supplement: Pea Protein Isolate, Rice Protein Concentrate, Hemp Protein
- Plant-based Protein, Then Whey Protein (Experimental): Performance tests/assessments will be conducted as baseline testing without plant-based protein, followed by four weeks of plant-based protein intervention consisting of one 70cc (32g) scoop of supplement provided within an hour after athletic practice, five days a week, for four weeks. For athletes with more than one practice a day, the supplement will be provided after the strength training session. The powder will be shaken with 8-12oz water. Performance measured at the end of 4 weeks.
  After a two-week washout period, they will undergo another performance evaluation and begin the same protein supplement regimen, but with a 70cc (32g) scoop of the whey protein supplement.
  Interventions: Dietary Supplement: Whey Protein Concentrate; Dietary Supplement: Pea Protein Isolate, Rice Protein Concentrate, Hemp Protein

INTERVENTIONS:
Dietary Supplement: Whey Protein Concentrate — whey-based protein powder 32g powder mixed with 8-12 oz water
  Other Names: True Nutrition Whey Protein Concentrate
  Arms: Plant-based Protein, Then Whey Protein; Whey Protein, Then Plant-based Protein
Dietary Supplement: Pea Protein Isolate, Rice Protein Concentrate, Hemp Protein — plant-based protein powder. 32g powder mixed with 8-12 oz water
  Other Names: True Nutrition Vegan Protein Optimizer Formula
  Arms: Plant-based Protein, Then Whey Protein; Whey Protein, Then Plant-based Protein

SUMMARY:
The objective of this study is to identify the prevalence of whey protein sensitivity in UIW athletes and to assess the effectiveness of 4-weeks of whey versus plant-based protein supplementation on athletic performance and recovery, specifically in those with whey sensitivity.

DETAILED DESCRIPTION:
Dependent t-tests and repeated measures analysis of variance (ANOVA) will offer comparative analyses between whey and plant protein conditions in subjects with and without whey sensitivity. Symptom questionnaires, perceived performance questionnaires, wearable fitness tracking data, and strength test results will be compared across all four conditions (baseline, washout, whey supplementation, and plant supplementation).

Related variables will be analyzed using GLM univariate, multivariate, and repeated measures. The overall multivariate Wilks' Lambda and Greenhouse-Geisser univariate p-levels will be reported. Differences among groups will be determined using Tukey's least significant differences (LSD) post hoc analyses.

ELIGIBILITY:
Inclusion Criteria:

* NCAA Division I collegiate athletes at the University of the Incarnate Word
* Must complete a medical history form
* Must be cleared by sports medicine staff for intercollegiate athletic participation

Exclusion Criteria:

* Individuals with a diagnosed food allergy, lactose intolerance, or inflammatory bowel disease (such as Chron's, Ulcerative Colitis, or Celiac Sprue)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Performance Questionnaire at 4 weeks | Baseline, 4 weeks, 6 weeks, 10 weeks
  subject assesses food sensitivity symptoms, perceived recovery after athletic event, and satisfaction with athletic performance.
Change from Baseline InBody Body Composition Test at 4 weeks | Baseline, 4 weeks, 6 weeks, 10 weeks
  Body composition assessed by subjects standing on bioelectrical impedance analysis scale that measures total body water, lean body mass, dy lean mass, body fat mass, and weight.
Change from Baseline Vertical Jump Test at 4 weeks | Baseline, 4 weeks, 6 weeks, 10 weeks
  The vertical jump measures explosive leg power and is an effective indirect measurement of athletic performance. The participant will utilize the Just Jump Mat to electronically assess vertical height.

SECONDARY OUTCOMES:
Number of Participants with Declining Measures | Baseline, 4 weeks, 6 weeks, 10 weeks
  The number of subjects whose self assessment, body composition, and vertical jump depreciate.
Number of Participants with Increasing Measures | Baseline, 4 weeks, 6 weeks, 10 weeks
  The number of subjects whose self assessment, body composition, and vertical jump improve.
Number of Athletes with Whey Sensitivity | Baseline
  Whey sensitivity assessed with IgG food sensitivity test, where small blood sample is collected from subject and IgG antibody level measured when introduced to whey.

CONTACTS AND LOCATIONS:
Overall Officials: Brittanie L Lockard, PhD, Principal Investigator — University of the Incarnate Word
Locations (1):
- The University of the Incarnate Word, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boirie Y, Dangin M, Gachon P, Vasson MP, Maubois JL, Beaufrere B. Slow and fast dietary proteins differently modulate postprandial protein accretion. Proc Natl Acad Sci U S A. 1997 Dec 23;94(26):14930-5. doi: 10.1073/pnas.94.26.14930. PMID 9405716
- [Background] Zopf Y, Baenkler HW, Silbermann A, Hahn EG, Raithel M. The differential diagnosis of food intolerance. Dtsch Arztebl Int. 2009 May;106(21):359-69; quiz 369-70; 4 p following 370. doi: 10.3238/arztebl.2009.0359. Epub 2009 May 22. PMID 19547751
- [Background] Anthoni S, Savilahti E, Rautelin H, Kolho KL. Milk protein IgG and IgA: the association with milk-induced gastrointestinal symptoms in adults. World J Gastroenterol. 2009 Oct 21;15(39):4915-8. doi: 10.3748/wjg.15.4915. PMID 19842221
- [Background] Malsagova, K, Stepanov, A, Sinitsyna, AA, Izotov, A, Klyuchnikov, MS, Kopylov, AT, and Kaysheva, AL. Determination of Specific IgG to Identify Possible Food Intolerance in Athletes Using ELISA. Data 6: 122, 2021.
- [Background] Stockton S, Breshears K, Baker DM. The Impact of a Food Elimination Diet on Collegiate Athletes' 300-meter Run Time and Concentration. Glob Adv Health Med. 2014 Nov;3(6):25-40. doi: 10.7453/gahmj.2014.046. PMID 25568830
- [Background] Lee LA, Burks AW. Food allergies: prevalence, molecular characterization, and treatment/prevention strategies. Annu Rev Nutr. 2006;26:539-65. doi: 10.1146/annurev.nutr.26.061505.111211. PMID 16602930
- [Background] Ozdemir O, Mete E, Catal F, Ozol D. Food intolerances and eosinophilic esophagitis in childhood. Dig Dis Sci. 2009 Jan;54(1):8-14. doi: 10.1007/s10620-008-0331-x. Epub 2008 Jul 2. PMID 18594978
- [Background] Zhou LM, Xu JY, Rao CP, Han S, Wan Z, Qin LQ. Effect of whey supplementation on circulating C-reactive protein: a meta-analysis of randomized controlled trials. Nutrients. 2015 Feb 9;7(2):1131-43. doi: 10.3390/nu7021131. PMID 25671415
- [Background] Benjamin J, Makharia G, Ahuja V, Anand Rajan KD, Kalaivani M, Gupta SD, Joshi YK. Glutamine and whey protein improve intestinal permeability and morphology in patients with Crohn's disease: a randomized controlled trial. Dig Dis Sci. 2012 Apr;57(4):1000-12. doi: 10.1007/s10620-011-1947-9. Epub 2011 Oct 26. PMID 22038507
- [Background] Antico A, Pagani M, Vescovi PP, Bonadonna P, Senna G. Food-specific IgG4 lack diagnostic value in adult patients with chronic urticaria and other suspected allergy skin symptoms. Int Arch Allergy Immunol. 2011;155(1):52-6. doi: 10.1159/000318736. Epub 2010 Nov 26. PMID 21109748
- [Background] Shakoor Z, AlFaifi A, AlAmro B, AlTawil LN, AlOhaly RY. Prevalence of IgG-mediated food intolerance among patients with allergic symptoms. Ann Saudi Med. 2016 Nov-Dec;36(6):386-390. doi: 10.5144/0256-4947.2016.386. PMID 27920409
- [Background] de Oliveira EP, Burini RC, Jeukendrup A. Gastrointestinal complaints during exercise: prevalence, etiology, and nutritional recommendations. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S79-85. doi: 10.1007/s40279-014-0153-2. PMID 24791919
- [Background] Lambert GP. Intestinal barrier dysfunction, endotoxemia, and gastrointestinal symptoms: the 'canary in the coal mine' during exercise-heat stress? Med Sport Sci. 2008;53:61-73. doi: 10.1159/000151550. PMID 19208999
- [Background] Marija, KV, Michalickova D, Dikic N, Stojmenovic T, Andjelkovic M, Nikolik I, Vukasinovic-Vesic M, and Malic T. Food elimination based on immunoglobulin G antibodies improves gastrointestinal discomfort symptoms and sport performance in professional athletes. Med Sport 70: 480-494, 2017.
- [Background] Jager R, Kerksick CM, Campbell BI, Cribb PJ, Wells SD, Skwiat TM, Purpura M, Ziegenfuss TN, Ferrando AA, Arent SM, Smith-Ryan AE, Stout JR, Arciero PJ, Ormsbee MJ, Taylor LW, Wilborn CD, Kalman DS, Kreider RB, Willoughby DS, Hoffman JR, Krzykowski JL, Antonio J. International Society of Sports Nutrition Position Stand: protein and exercise. J Int Soc Sports Nutr. 2017 Jun 20;14:20. doi: 10.1186/s12970-017-0177-8. eCollection 2017. PMID 28642676
- [Background] Protein Supplements Market Size Report, 2021-2030. 2022, 2022.
- [Background] Gorissen SHM, Crombag JJR, Senden JMG, Waterval WAH, Bierau J, Verdijk LB, van Loon LJC. Protein content and amino acid composition of commercially available plant-based protein isolates. Amino Acids. 2018 Dec;50(12):1685-1695. doi: 10.1007/s00726-018-2640-5. Epub 2018 Aug 30. PMID 30167963
- [Background] Lim MT, Pan BJ, Toh DWK, Sutanto CN, Kim JE. Animal Protein versus Plant Protein in Supporting Lean Mass and Muscle Strength: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2021 Feb 18;13(2):661. doi: 10.3390/nu13020661. PMID 33670701
- [Background] US BioTek Laboratories, L. See All Our Tests | US BioTek Laboratories, 2022.
- [Background] Hooper SL, Mackinnon LT. Monitoring overtraining in athletes. Recommendations. Sports Med. 1995 Nov;20(5):321-7. doi: 10.2165/00007256-199520050-00003. No abstract available. PMID 8571005
- [Background] Laurent CM, Green JM, Bishop PA, Sjokvist J, Schumacker RE, Richardson MT, Curtner-Smith M. A practical approach to monitoring recovery: development of a perceived recovery status scale. J Strength Cond Res. 2011 Mar;25(3):620-8. doi: 10.1519/JSC.0b013e3181c69ec6. PMID 20581704
- [Background] Bukhari, FK, Fahd, S, Tahira, R, and Yaseen, M. Impact of Sports Anxiety on Sports Performance of Players. Pakistan Journal of Humanities and Social Sciences 9, 2021.
- [Background] Ling CH, de Craen AJ, Slagboom PE, Gunn DA, Stokkel MP, Westendorp RG, Maier AB. Accuracy of direct segmental multi-frequency bioimpedance analysis in the assessment of total body and segmental body composition in middle-aged adult population. Clin Nutr. 2011 Oct;30(5):610-5. doi: 10.1016/j.clnu.2011.04.001. Epub 2011 May 8. PMID 21555168
- [Background] Klavora, P. Vertical-jump Tests: A Critical Review. Strength and Conditioning Journal. October 2000 22:5.
- [Background] Jenni. WHOOP Strain. Retrieved April 22, 2022, from https://support.whoop.com/hc/en-us/articles/360019453214-WHOOP-Strain
- [Background] Van Deusen, M. Heart Rate Variability | The Ultimate Guide to HRV. 2022, 2021.
- [Background] Berryhill S, Morton CJ, Dean A, Berryhill A, Provencio-Dean N, Patel SI, Estep L, Combs D, Mashaqi S, Gerald LB, Krishnan JA, Parthasarathy S. Effect of wearables on sleep in healthy individuals: a randomized crossover trial and validation study. J Clin Sleep Med. 2020 May 15;16(5):775-783. doi: 10.5664/jcsm.8356. Epub 2020 Feb 11. PMID 32043961
- [Background] Garza B, Ege T, Ramos S, Lockard B. Comparison of Actual versus Recommended Intake of Collegiate Athletes Across Gender and Season at a Small Division I University. International Journal of Exercise Science: Conference Proceedings, 2022.